CLINICAL TRIAL: NCT06161701
Title: A Study on the Influencing Factors of Glucocorticoid Induced Elevated Blood Glucose in Nephrotic Patients
Brief Title: Steroid Diabetes in Patients With Kidney Disease
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Provincial People's Hospital (Other)
Collaborators: The Third Affiliated Hospital of Wenzhou Medical University (Other); The First People's Hospital of Xiaoshan District, Hangzhou City (Unknown); The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other); Nanxun District People's Hospital of Huzhou City，China (Unknown); Wenling Traditional Chinese Medicine Hospital (Unknown); Affiliated Hospital of Jiaxing University (Other); Taizhou Hospital (Other); The First People's Hospital of Chun'an (Unknown)
Responsible Party: Sponsor
Other Study IDs: KT20220083
Record Dates: First submitted 2023-08-22; First posted 2023-12-08 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Nephrotic Syndrome
Keywords: steroid diabetes
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Blood glucose management in patients with kidney disease after using glucocorticoids: Blood glucose monitoring for kidney disease patients after taking glucocorticoids
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
If steroid diabetes is not recognized in time, it will cause irreversible damage to the body. Nephropathy patients are more likely to have steroid diabetes ,the incidence rate up to 25%,due to hypoalbuminemia, high-dose hormone and other reasons, so they need to be closely followed up, identified and intervened in time.

DETAILED DESCRIPTION:
1. Patients with nephrosis who had taken glucocorticoid for the first time were followed up, and those who had diabetes themselves were excluded.
2. Regularly follow up and record information on glucocorticoid medication, medications that have an impact on blood sugar, fasting blood sugar, 2-hour postprandial blood sugar, and glycated hemoglobin.
3. Notify relevant doctors of any cases of elevated blood sugar.
4. The total follow-up time is 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who need to use glucocorticoids due to the following diseases: nephrotic syndrome, Immunoglobulin A nephropathy, membranous nephropathy, Anti-neutrophil cytoplasmic antibodies (ANCA)-associated vasculitis (AAV), systemic lupus erythematosus；
2. Initial daily dose of glucocorticoids greater than or equal to 10mg of prednisolone；

Exclusion Criteria:

1. Patients with diabetes；
2. Those who are unable to communicate through language；
3. Uremic patients；
4. Unable to perform blood glucose monitoring and follow-up as required；
5. Those who have used glucocorticoids within the past 3 months and have accumulated a dose of 10mg or more of prednisone；
6. Participated in other clinical studies。

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient or inpatient kidney disease patients seeking treatment at any research hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of steroid diabetes in nephrotic patients after glucocorticoid use | If the use of glucocorticoids exceeds one year, observe for one year; If the usage time is less than one year, observe 3 months after discontinuation of medication.
  steroid diabetes is defined as the absence of diabetes in the past, which occurs after the use of glucocorticoid:
  1. Typical symptoms accompanied by any of the following:
     Fasting blood glucose ≥ 7.0mmol/L or random blood glucose ≥ 11.1mmol/L or plus OGTT 2-hour blood glucose ≥ 11.1mmol/L; Or glycated hemoglobin is greater than or equal to 6.5%;
  2. If there are no typical symptoms, then it needs to meet any two or more of the above results;
  The incidence of steroid diabetes is defined as the number of patients diagnosed with steroid diabetes after glucocorticoid use/the number of patients enrolled * 100%

SECONDARY OUTCOMES:
Cumulative use time of glucocorticoid, cumulative dose of glucocorticoid and drugs that may affect blood glucose in combination with steroid diabetes | Time from enrollment to steroid diabetes happens
  The cumulative use time of glucocorticoid refers to the time from regular use of glucocorticoid to steroid diabetes;
  The cumulative dose of glucocorticoid refers to the cumulative dose of glucocorticoid from the time of regular use of glucocorticoid to the time of occurrence of steroid diabetes, calculated by prednisone;
  Medications that may affect blood sugar in combination therapy: Tacrolimus, cyclosporine, hydrochlorothiazide β- Receptor blockers, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolan Ye, master, Study Director — Zhejiang Provincial People's Hospital
Locations (1):
- Zhejiang provincial people's hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
One year after the completion of the study, for researchers who do require relevant data, the basic characteristics of enrolled cases and the development and changes of blood sugar can be provided by email.